CLINICAL TRIAL: NCT03426488
Title: Northern Sweden Health and Disease Study
Acronym: NSHDS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Responsible Party: Sponsor
Other Study IDs: Umu
Record Dates: First submitted 2017-12-18; First posted 2018-02-08 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2017-12

CONDITIONS: Cardiovascular Diseases; Cancer; Neurodegenerative Diseases; Respiratory Disease; Infection
MeSH Terms: conditions — Cardiovascular Diseases; Neoplasms; Neurodegenerative Diseases; Respiration Disorders; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The blood samples consist primarily of EDTA and heparin blood samples divided into plasma, erythrocyte concentrate and buffy coat and for a certain percentage, the DNA is extracted.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Västerbotten Intervention Programme: The cohort is population-based and consists of blood and data from primarily 40, 50 and 60 year olds, taken every year in this age group in connection with the Västerbotten health surveys from 1985 - present.
  The blood samples consist primarily of EDTA and heparin blood samples divided into plasma, erythrocyte concentrate and buffy coat and for a certain percentage, the DNA is extracted.
  The database NSDD (Northern Sweden Diet Database) consists of survey data from VIP concerning nutritional factors.
  A large part is fasting samples.
  Individuals: 105,700 Individuals with repeated samples: 40,700 Sampling occasions: 156,300
  Interventions: Behavioral: VIP - Västerbotten Intervention Programme
- Mammography Screening Project: Samples and data are collected in connection with mammography screenings 1995-2006. The blood samples consist primarily of EDTA and heparin blood samples divided into plasma, erythrocyte concentrate and buffy coat, and for a certain percentage, the DNA is also extracted. The cohort consists of women, 18-82 years old (95% between 48 and 70 years old).
  Survey data can be linked to the blood samples.
  Individuals: 28,800 Individuals with repeated samples: 14,600 Sampling occasions: 54,000
- The Northern Swedish MONICA Project: The MONICA study is a longitudinal population-based database for research in cardiovascular disease and diabetes. Since 1985, seven screenings has been performed (1986, 1990, 1994, 1999, 2004, 2009 and 2014) of a randomized selection of the population in the counties of Västerbotten and Norrbotten in Northern Sweden.
  Individuals: 11,800 Individuals with repeated samples: 3,500 Sampling occasions: 15,300 (March 2015)

INTERVENTIONS:
Behavioral: VIP - Västerbotten Intervention Programme — Intervention on CVD (cardiovascular disease) and diabetes
  Groups: Västerbotten Intervention Programme

SUMMARY:
NSHDS (Northern Sweden Health and Disease Study) is an umbrella term for a prospective biobank with related survey data. The sample collection consists of three subcohorts, Västerbotten Intervention Programme (VIP), Mammography Screening Project (MA) and MONICA (MONItoring of Trends and Determinants in CArdiovascular Disease). The blood samples are stored at the Northern Sweden Biobank.

DETAILED DESCRIPTION:
The overall aim of the NSHDS is to support frontline research with particular emphasis on improving diagnostic tools for clinical use, as well as finding early markers of disease, using the blood samples, tissue and associated health data from the NSHDS. Furthermore, basic research regarding risk factors as well as pathogenetic pathways are promoted.

The prospective blood samples and related survey data can be linked to national registries for health outcomes such as cancer diagnosis for which there is a near 100% completeness of the data.

VIP - VÄSTERBOTTEN INTERVENTION PROGRAMME The VIP is a long-term project intended for health promotion of the population of the county of Västerbotten (approximately 254,000 inhabitants). All individuals 40, 50, and 60 years of age in the county are invited for screening. They are asked to complete a questionnaire concerning various lifestyle factors, including diet, and to donate a blood sample to be frozen for later research purposes. The cohort is population-based and the inclusion of individuals started 1985 and is ongoing. The participation rate has ranged between 48 and 67% of the population. But a large number has not been invited for screening. Among those invited the participation rate has been very high. The material is population based.

The blood samples consist primarily of EDTA (ethylenediaminetetraacetic acid) and heparin blood samples divided into plasma, erythrocyte concentrate and buffy coat. Questionnaire data are linked to blood samples.

The majority of samples are fasting samples. Number of individuals: 103,100 Individuals with repeated samples: 43,500 Sampling occasions: 151,200 (October 2016)

MA - MAMMOGRAPHY SCREENING PROJECT

Samples and data are collected in connection with mammography screenings 1995-2006. The blood samples consist primarily of EDTA and heparin blood samples divided into plasma, erythrocyte concentrate and buffy coat, and for a certain percentage, the DNA is also extracted. The cohort consists of women, 18-82 years old (95% between 48 and 70 years old).

Survey data can be linked to the blood samples.

Individuals: 28,800 Individuals with repeated samples: 14,600 Sampling occasions: 54,000

THE MONICA STUDY

The MONICA study is a longitudinal population-based database for research in cardiovascular disease and diabetes. Since 1985, seven screenings has been performed (1986, 1990, 1994, 1999, 2004, 2009 and 2014) of a randomized selection of the population in the counties of Västerbotten and Norrbotten in Northern Sweden.

Individuals: 11,800 Individuals with repeated samples: 3,500 Sampling occasions: 15,300

This registration will only cover blood sampling (screenings since 1990) and dietary data (optional MONICA study, screenings since 1986) as a part of the National Environmental Biobank. The participation rates have been 69-81%.

A separate registration is expected for the basic MONICA study.

ELIGIBILITY:
Inclusion Criteria:

* Residents in Northern Sweden

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Given before
Sampling Method: Probability Sample
Enrollment: 120000 (Estimated)
Dates: Start 1986-01 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Number of deaths | Follow up at least 20 years
Numbers of incident cases of disease. | Follow up at least 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Göran Hallmans, MD PhD, Principal Investigator — Umeå University
Locations (1):
- Umeå University, Umeå, Västerbotten County, Sweden

IPD SHARING:
Plan to Share IPD: No